CLINICAL TRIAL: NCT01722799
Title: PROSPECTIVE RANDOMIZED TRIAL Multicentric Study to Evaluate the Treatment and the Efficiency of Paclitaxel-coated Balloon IN.PACT FALCON ® in Small-vessel Coronary Stenosis.
Brief Title: Randomized Trial of Coronary Angioplasty for de Novo Lesions in sMall vesSElS With Drug Eluting Balloon.
Acronym: RAMSES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andres Iñiguez Romo, MD, PhD (Other Government)
Responsible Party: Sponsor-Investigator, Andres Iñiguez Romo, MD, PhD, Dr. Andres Iñiguez Romo, Hospital de Meixoeiro
Organization: Hospital de Meixoeiro (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEIX-STENT-001; RAMSES-DEB (Other Grant/Funding Number: BIOMEDICAL FUNDATION VIGO)
Record Dates: First submitted 2012-09-25; First posted 2012-11-07 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Coronary Disease
Keywords: angioplasty; Percutaneous Transluminal Coronary Angioplasty; Drug elluting Balloon; Coronary Balloon; Dilatation
MeSH Terms: conditions — Coronary Disease; Dilatation, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug elluting Balloon (DEB) (Experimental): Is a coronary dilating device with Paclitaxel ® drug delivery, for dilatation and provisional spot bare metal stenting (BMS).
  Interventions: Device: Drug elluting Balloon (DEB)
- Drug elluting coronary stent (DES) (Active Comparator): The Resolute Integrity Zotarolimus-Eluting Coronary Stent System is indicated for improving coronary luminal diameters in patients, including those with diabetes mellitus, with symptomatic ischemic heart disease due to de novo lesions of length ≤ 27 mm in native coronary arteries with reference vessel diameters of 2.25 mm to 4.20 mm.
  Interventions: Device: Drug elluting coronary stent (DES)

INTERVENTIONS:
Device: Drug elluting Balloon (DEB) — Percutaneous transluminal coronary angioplasty with drug elluting ballon and Bare metal stent for rescue.
  Other Names: IN.PACT™ Falcon paclitaxel eluting balloon.
  Arms: Drug elluting Balloon (DEB)
Device: Drug elluting coronary stent (DES) — Percutaneous transluminal coronary angioplasty (PTCA) with stent
  Other Names: Resolute integrity™ zotarolimus drug coronary stent
  Arms: Drug elluting coronary stent (DES)

SUMMARY:
Significant lesions in small coronary arteries are frequently found (35%-50%) in patients with coronary artery disease. Independently of the type of coronary angioplasty the restenosis and the need for repeat revascularization remains the main limitation, representing a challenging problem even in the DES (drug eluting stent) era. Recently has been developed drug eluting balloons (DEBs), which have been successfully tested in small series on in-stent restenosis, but few evidence is available in the context of small vessels disease.

The current study has been designed to know, in one hand, the clinical efficacy of the Drug elluting balloon IN.PACT FALCON and, in other hand, the effectiveness, and the cost-effectiveness incremental analysis of DEBs (IN.PACT FALCON vs. DES ( RESOLUTE INTEGRITY) in patients with de novo lesions in small vessels.

DETAILED DESCRIPTION:
Recent studies have reported the efficacy of the local application of paclitaxel ® inhibiting neointimal proliferation, and thus the limitation of restenosis, which has led to the conception and development of drug-coated balloon or "Drug Eluting Balloons" (DEB), releasing the antiproliferative drug at the time of expansion. Initially they were applied in the treatment of in-stent restenosis. However, DEB may represent a therapeutic alternative in other contexts where anatomo-clinical uses are not always therapeutic percutaneous coronary revascularization with stent implantation, as is the case of coronary lesions located in small vessels.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18, informed consent.
2. Evidence of CAD with severe de novo lesion in the native coronary arteries ( ≥70% stenosis by visual estimation or >50% by CT scan); affecting
3. Vessels between 2,25 and 2,75 mm diameter and
4. The length of the coronary stenosis ≤25 mm
5. Patient informed consent form signed.

Exclusion Criteria:

1. Lesion in coronary left main ,
2. Chronic total occlusions,
3. Lesions at bifurcation,
4. Severe calcified lesions,
5. Lesions in aorto-coronary saphenous veins or arterial grafts,
6. Acute Myocardial Infarction during 48 hours before the procedure,
7. Severe renal dysfunction,
8. Hypersensibility, allergy or contraindication of medication: acetylsalicylic acid, clopidogrel, ticlopidine, heparin, paclitaxel,
9. Allergy to contrast media,
10. Life expectancy less than 1 year,
11. 1 year FU not guaranteed,
12. Being participating in another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
Compare the clinical efficacy measured by target vessel failure of DEB IN.PACT FALCON DEB versus the resolute integrity stent (DES). | The efficacy will be evaluated at 1 year.
  Target vessel failure (TVF) is define as any revascularization motivated due to myocardial infarction (with or without Q wave) or cardiac death related to the target vessel.
Compare the clinical security measured by the incidence MACE of DEB IN.PACT FALCON DEB versus the resolute integrity stent (DES). | The security will be evaluated at one month, sixth month and one year
  Rate of major adverse cardiac events (MACE) at 30 days, 6 months and one year. MACE was defined as cardiac death, myocardial infarction (MI) (with or without Q-wave), need for repeat revascularization of the treated vessel (surgical or repeat PCI) or occlusion of the treated lesion.

SECONDARY OUTCOMES:
Compare the efficiency of DEBs versus DES. in terms of cost effectiveness (cost per adverse event-death avoided) and cost-utility ( cost per quality adjusted life year) in patients with de novo lesions in small vessels. | The efficiency will be evaluated at first month, 6 month and 1 year.
  In order to perform a cost-utility analysis, years of quality-adjusted life (QALY) gained will be measured using the quality of life questionnaire EuroQoL five dimensions (EQ-5D) and a visual scale at baseline, one month and 12 months.
Compare the direct cost, indirect costs and total costs of DEBs versus DES in patients with de novo lesions in small vessels. | This outcome will be evaluated at first month, 6 month and 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Iñiguez Romo, MD,PHD, Principal Investigator — Hospital Universitario Alvaro Cunqueiro; Victor A. Jimenez Diaz, MSC, Principal Investigator — Hospital Universitario Alvaro Cunqueiro; Pablo M Juan Salvadores, Pharma; MPH, Study Director — Hospital Universitario Alvaro Cunqueiro; Jose M. Hernández García., MD, Principal Investigator — Hospital Virgen de la Victoria; Eduardo Molina Navarro, MD, Principal Investigator — Hospital Virgen de las Nieves; Francisco Bosa Ojeda, MD, Principal Investigator — Complejo Hospitalario Universitario de Canarias; Armando Pérez de Prado, MD, Principal Investigator — Hospital Universitario de Leon; Fernando Lozano Ruiz-Poveda, MD, Principal Investigator — Hospital Universitario de Ciudad Real; Cristobal A. Urbano Carrillo, Principal Investigator — Hospital Clínico Universitario Carlos Haya
Locations (1):
- Hospital Universitario Álvaro Cunqueiro, Vigo, Pontevedra, Spain

REFERENCES:
- [Result] Tepe G, Schmitmeier S, Speck U, Schnorr B, Kelsch B, Scheller B. Advances on drug-coated balloons. J Cardiovasc Surg (Torino). 2010 Feb;51(1):125-43. PMID 20081769
- [Result] Schnorr B, Kelsch B, Cremers B, Clever YP, Speck U, Scheller B. Paclitaxel-coated balloons - Survey of preclinical data. Minerva Cardioangiol. 2010 Oct;58(5):567-82. PMID 20948503
- [Result] Unverdorben M, Vallbracht C, Cremers B, Heuer H, Hengstenberg C, Maikowski C, Werner GS, Antoni D, Kleber FX, Bocksch W, Leschke M, Ackermann H, Boxberger M, Speck U, Degenhardt R, Scheller B. Paclitaxel-coated balloon catheter versus paclitaxel-coated stent for the treatment of coronary in-stent restenosis. Circulation. 2009 Jun 16;119(23):2986-94. doi: 10.1161/CIRCULATIONAHA.108.839282. Epub 2009 Jun 1. PMID 19487593
- See also: Web Page from Cardiology department.Hospital Meixoeiro. — http://www.cardiologia-vigo.com